CLINICAL TRIAL: NCT05120206
Title: Outcomes of Periodontal Therapy in Smokers and Non-smokers With Chronic Periodontitis
Brief Title: The Impact of Cigarette Smoking on Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 94605
Record Dates: First submitted 2021-10-05; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis; Cigarette Smoking
MeSH Terms: conditions — Periodontitis; Cigarette Smoking | interventions — Educational Status; Oral Hygiene; Gingivectomy; chlorhexidine gluconate; Chlorhexidine; halofantrine

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cigarette smokers with periodontitis (Active Comparator): Periodontal therapy in cigarette smokers
  Interventions: Procedure: Non-surgical periodontal therapy: motivation and instruction in oral hygiene, debridement using handinstrumentation (Hu-Firedy,Chicago, IL, USA;and American Eagle Instruments,Missoula, MT,USA).
- Non-smokers with periodontitis (Active Comparator): Periodontal therapy in non-smokers
  Interventions: Procedure: Non-surgical periodontal therapy: motivation and instruction in oral hygiene, debridement using handinstrumentation (Hu-Firedy,Chicago, IL, USA;and American Eagle Instruments,Missoula, MT,USA).

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy: motivation and instruction in oral hygiene, debridement using handinstrumentation (Hu-Firedy,Chicago, IL, USA;and American Eagle Instruments,Missoula, MT,USA). — Non-surgical and surgical periodontal therapy in cigarette smokers and non-smokers
  Other Names: Periodontal surgery: periodontal flap and gingivectomy with postoperative rinse with 0.2% chlorhexidine gluconate (Corsodyl, GlaxoSmithKline, London, UK).

SUMMARY:
Periodontitis patients, 40 cigarette smokers and 40 non-smokers (defined by cotinine measures in serum), were recruited to this double arm prospective cohort study. Data were collected 3 months following non-surgical and surgical periodontal treatment, and following 12 months with supportive periodontal therapy. Data collected were clinical attachment level, probing depth, bleeding on probing,oral bacteria, serum, blood (PAXgeneBlood), and gingival crevicular fluid.

DETAILED DESCRIPTION:
The overall aim of this work was to study clinical outcomes of active and supportive periodontal therapy in smokers and non-smokers with chronic periodontitis at patient, tooth, and site level. Moreover, to compare the periopathogenic microflora and inflammatory markers in gingival crevicular fluid and in blood in smokers and non-smokers following therapy.

Eighty patients, 40 smokers and 40 non-smokers, with moderate to severe chronic periodontitis were included in this prospective cohort study and treated non-surgically and surgically, and then followed-up in a supportive periodontal therapy program for 12 months. Smoking status was validated measuring serum cotinine levels at pre-treatment and 12 months following supportive periodontal therapy.

Clinical measurements included full mouth recordings of clinical attachment level, probing depth, bleeding on probing, and plaque index at pre-treatment and following active and supportive periodontal therapy. At the same timepoints, subgingival plaque samples of 20 subgingival periopathogenic bacterial species were analysed using checkerboard DNA-DNA hybridization. Blood samples (PAXgeneBlood), serum, gingval crevicular fluid were also collected at the three timepoints.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* age 35-75 years
* diagnosed with chronic periodontitis
* at least four non-adjacent teeth with proximal sites with a PD ≥6 mm and clinical attachment loss ≥5 mm with BoP and no radiographic signs of apical pathology.
* either smokers (>10 cigarettes per day for at least 5 years) or non-smokers (never smoked or not within the last 5 years).

Exclusion Criteria:

* subjects who presented with any current medical condition or used medications known to affect periodontal healing
* incorrectly reported smoking status
* use of antibiotics within 6 months of the study
* received subgingival scaling within 6 months of the study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
PD ≥5 mm with BoP | 24 months
  Corrected for clustering within patients, teeth, and sites over time, was the unit of the analysis and PD ≥5 mm with BoP was the outcome (dependent variable) dichotomized as present (1) or absent (0).

SECONDARY OUTCOMES:
Teeth present | 24 months
  Number of teeth
Clinical periodontal attachmentloss | 24 months
  Clinical attachment loss in mm
Periodontal pocket depth | 24 months
  Probing depth in mm
Bleeding at site level | 24 months
  Bleeding on probing (yes or no)
Bleeding at patient level | 24 months
  Bleeding index in percentage (%)
Plaque at patient level | 24 months
  Plaque index in percentage (%)
Amount of periopathogenic bacteria | 24 months
  Subgingival plaque samples of 20 subgingival periopathogenic bacterial species were analysed using checkerboard DNA-DNA hybridization.
Inflammatory gingival crevicular fluid markers (proteins) | 24 months
  Concentrations of gingival crevicular fluid biomarkers measured in pg/mLwere analysed using multiplex and singleplex micro-bed immunoassays.
Serum proteins | 24 months
  Concentration of inflammatory serum markers measured in pg/ɥL determined using multiplex kit Bio-Plex Human ProTM Assay.
Gene expression in blood | 24 months
  Inflammatory gene (RNA) expression levels is estimated by counting the reads that map to genes or exones using the the RPKM (Reads per Kilobases per Million reads) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar F. Bunæs, PhD, Principal Investigator — Department of Clinical Dentistry - periodontics, University of Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bunaes DF, Lie SA, Enersen M, Aastrom AN, Mustafa K, Leknes KN. Site-specific treatment outcome in smokers following non-surgical and surgical periodontal therapy. J Clin Periodontol. 2015 Oct;42(10):933-42. doi: 10.1111/jcpe.12462. Epub 2015 Oct 28. PMID 26407817
- [Result] Bunaes DF, Mustafa M, Mohamed HG, Lie SA, Leknes KN. The effect of smoking on inflammatory and bone remodeling markers in gingival crevicular fluid and subgingival microbiota following periodontal therapy. J Periodontal Res. 2017 Aug;52(4):713-724. doi: 10.1111/jre.12438. Epub 2017 Mar 17. PMID 28306142